CLINICAL TRIAL: NCT05927584
Title: Local Excision for Organ Preservation in Early REctal Cancer With No Adjuvant Treatment (LORENA Trial).
Brief Title: Local Excision for Organ Preservation in Early REctal Cancer With No Adjuvant Treatment
Acronym: LORENA
Status: Recruiting | Type: Observational
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Collaborators: Hospital Alemão Oswaldo Cruz (Other); Hospital Universitario La Fe (Other); Complejo Hospitalario Universitario de Vigo (Other)
Responsible Party: Sponsor
Other Study IDs: HUP-23/5216
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Rectal Cancer; Rectum Neoplasm
Keywords: Early rectal cancer; Local excision; Total Mesorectal Excision; Organ preservation
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: None Retained — Rectal cancer transanal local excision specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Local excision: * Patients older than 18 years
  * Diagnosis of rectal cancer
  * Inferior edge of the tumour not further than 2 cm above the anorectal ring
  * Clinical TNM staging T1N0M0
  Interventions: Procedure: Transanal local excision

INTERVENTIONS:
Procedure: Transanal local excision — Transanal full thickness local excision

SUMMARY:
Rectal cancer is one of the most frequent malignant tumors nowadays. There are several possible treatment options including chemotherapy, radiotherapy and surgery. Surgery for early stage rectal cancer can be either a radical surgery (RS) or a local excision (LE).

A radical surgery removes the rectum including the tumor and the lymph nodes through which it spreads, improving survival but with a possible impact in the patients quality of life (QoL). A local excision only removes the tumor and a safety margin of healthy rectum. This has the potential to avoid the possible complications and QoL decrease. However there are some complications after a LE and also poor prognostic factors inherent to the tumor biology that can lead the surgical team to perform a RS after LE with worse outcomes. These are impossible to know before the procedure.

The goal of this registry is to determine the frequency of these poor prognostic biological factors and complications in patients undergoing LE for early rectal cancer.

The main question it aims to answer are:

• How frequently does LE allow for rectum preservation?

Participants will undergo LE for early rectal cancer when it is considered the best treatment by their surgeons according to their expertise and protocols. Patients will follow the standard treatment that would be given to them, and the biological prognostic factors and the appearance of complications will be recorded.

DETAILED DESCRIPTION:
Registry´s main hypothesis:

Exclusive LE is insufficient for in situ rectum preservation in cT1N0M0 extraperitoneal rectal adenocarcinoma in ≥20% of the patients treated with this approach in real everyday´s clinical practice.

A database will be design recording demographics, tumor details, type of intervention, complications, histological details and further necessity of treatments and rectal preservation along time. It will be hosted online through the REDCap system.

Data entry will be done baseline, after surgical procedure, and at different follow-up periods, at 30 postoperative day and at 6, 12, 18, 24 and 36 months after surgical intervention.

Sample size calculation:

Previous evidence states that most patients would be willing to assume a recurrence risk of 20% (IQR 10-35%) in locally advanced rectal cancer after chemo-radiotherapy in order to join the watch and wait strategy for organ preservation. In the project the investigators propose a salvage TME rate of less than 20% at three years to be acceptable. With this approach, accepting a risk α of 0.05 and a risk β of 0.2, a two-tailed test would require a total of 145 patients to identify a difference of 0.1 units. A proportion in the reference group of 0.2 and a loss rate of 5% has been estimated.

Clinical variables

Clinical and demographic data will be collected from each patient, using their computerised clinical history, and a data collection notebook will be prepared.

* Centre code: Each participating centre will receive a unique code that will be the first variable in the database in order to identify the participation of each centre in the study.
* Patient code: Each patient included in each centre will receive a consecutive numerical code to identify the different cases registered in the study.
* Demographic variables: Sex, date of birth, weight (kg), height (cm).
* Comorbidities and cardiovascular risk factors: ASA classification, diabetes mellitus, hypertension, dyslipidaemia, smoking, heart disease, immunosuppression.
* Preoperative laboratory values: haemoglobin (mg/dl), albumin (mg/dl), carcinoembryonic antigen (mg/dl).
* Preoperative clinical staging: Tests performed (MRI, endoanal ultrasound, endoscopic techniques), distance of the tumour to the ano-rectal ridge, distance of the tumour to the external anal margin, tumour size (cranial-caudal axis), percentage of rectal circumference occupation (<25%, 25-50%, >50%).
* Operative data: Date of resection, resection approach (endoscopic vs. surgical), transanal resection devices (TEM, TEO, TAMIS, Robot-TAMIS), technique used (local full-wall resection vs. submucosal dissection), intraoperative complications (bleeding, vaginal perforation, tumour perforation/rupture), medical complications).
* Postoperative complications: Clavien-Dindo classification, wound dehiscence, surgical site infection, bleeding.
* Pathological data: pT classification, histological grade, circumferential margins, vascular, lymphatic and perineural infiltration, micron infiltration of submucosa and tumour budding.
* Need to complete treatment: Reason (local resection complication, high risk factors, inadequate surgical margins, piecemeal resection, local recurrence, final pathological staging greater than pT1), radical surgery (dichotomous), technique used (total mesorectal excision, abdominoperineal amputation of rectum), time from local excision to radical surgery (date), stoma preparation (dichotomous), type of stoma (ileostomy vs. Colostomy, temporary vs. definitive), transit reconstruction within the study period (in temporary stomas), adjuvant radiotherapy, adjuvant radio-chemotherapy,
* Follow-up: complications recorded prospectively at 60 days by means of periodic visits to the coloproctology clinic, with the end of follow-up for the patient within the study being the annual check-up. The number of consultations during the first year, recurrence (indicating date and management) and death will be assessed. Oncological follow-up will be carried out with control of tumour markers (CEA), control imaging tests (CAT scan associated with PET/CT in the case of recurrence), and selected biopsies according to the results.

Statistical method:

The data obtained from each patient will be entered into a database and the analysis will be performed with a statistical programme Stata 13.1 (StataCorp, Texas, USA).

A descriptive analysis of demographic and clinical variables will be performed. Categorical variables will be presented as percentages and frequencies. Qualitative variables will be presented as percentages and frequencies. Quantitative variables will be described as mean and standard deviation (SD) if they follow a normal distribution or as median and interquartile range (IQR), in case of skewness.

The association between the variables collected and the target variables of the study will be performed by Pearson's Chi-square test or Fisher's exact test, as appropriate, in the case of categorical variables and, for continuous variables, by Student's t-test for independent samples or Mann-Whitney U-test, respectively, depending on whether or not their distribution conforms to the normal distribution.

Overall survival, disease-free survival, local recurrence-free survival and overall mesorectal resection-free survival will be estimated using the Kaplan-Meier method and the Cox proportional hazards model. Patients lost to follow-up will be censored.

Chronogram and study´s stages:

* March - September, 2023: Study´s protocol design and approval by the promoter center´s local ethics committee. Recruitment period for other participant centers.
* October,- December 2023: Unique registry database design in the REDCap platform.
* January 2024 - December 2024: Recruitment of the necessary cases according to the sample size calculation.
* January - December 2025: 1-year follow-up of patients included in the study.
* January - April 2026: Interim analysis after the first year of oncologic follow-up for assessment of the primary endpoint of the study (organ preservation with exclusive local resection) as well as some of the secondary endpoints.
* December 2027: Follow-up period to complete the study at 3 years.

Ethical and legal aspects:

The investigation will be conducted according to the 2013 Fortaleza´s update of the the Helsinki Declaration, and to each participant´s country law.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 years or older.
* Histologic proof of infiltrating rectal adenocarcinoma. or
* Preoperative biopsy compatible with rectal adenoma or intramucous adenocarcinoma with endoscopic or radiological suspicion of infiltrating adenocarcinoma.

  1. Endoscopic criteria: Kudo´s crypt pattern of V or higher, despite non confirmatory preoperative histology. endoscópicos: patrón de criptas V o superior según la clasificación de Kudo, que define lesiones infiltrantes, a pesar de que la histología preoperatoria no sea confirmatoria .
  2. Ultrasonographic criteria: hipoecogenic rectal tumor invading the intermediate hyperecogenic layer (submucosal), but does not infiltrate the hypoecogenic outer layer (muscularis propia).
  3. Radiological criterio in MR: tumor invades the submucosal layer without infiltration of the rectal muscularis propia. The usual low signal submucosal image is substituted with an aberrant signal, meaning the loss of the zebra pattern in a normal rectal wall.
* Rectal neoplasm with an inferior limit no further than 2cm proximal to the anorectal verge, both in digital rectal examination and in radiology examinations, ideally magnetic resonance (MR).
* Rectal neoplasms up to 3 cm of major diameter.
* Clinical preoperative staging of cT1N0M0, based on endoscopy, MR, +/- endorectal ultrasound.
* Cases in which LE as exclusive treatment with curative intent is prescribed after MDT discusión, regardless of the approach both via flexible endoscopy and transanal endoscopic microsurgery and its variations.
* Neoplasms with low risk histologic criteria known preoperatively or lack of information regarding this aspect:

  1. Submucosal infiltration of less than 1000µm (sm1 in the Kikuchi classification) .
  2. Tumor budding absent.
  3. En bloc resection in patients with a previous endoscopic resection.
  4. Vascular, lymphatic and perineural invasión absent.
  5. Low histologic grade.

Exclusion Criteria:

* Patients younger than 18 years old.
* Rectal neoplasms different from adenocarcinoma.
* Neoplasms in which the inferior edge is farther than 2cm proximal to the anorectal verge in the preoperative MR.
* Any other clinical stage other than cT1N0M0 (any T>1, N+, or M+).
* Neoplasms larger than 3cm.
* Preoperatively demonstration of PPHF:

  1. Submucosal infiltration deeper than 1000µm (sm2 and sm3 in the Kikuchi classification)
  2. Tumor budding present.
  3. Piecemeal resection in cases with previous endoscopic resection.
  4. Vascular, lymphatic and perineural invasión presence.
  5. High histologic grade.
* Any patient with planned systemic treatment with RTQT combined with the LE after MDT discusión, regardless of the preoperative clinical or postoperative pathological stage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with early stage rectal cancer, meaning clinical TNM staging cT1N0M0, programmed to receive Local Excision as an exclusive therapy according to each center´s standard practice.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Success rate | 36 months
  Rate of patients with no need of Total Mesorectal Excision after follow-up

SECONDARY OUTCOMES:
Morbidity rate | 2 months
  Postoperative complication rate, description, and severity according to Clavien Dindo classification
Radicality of resection | 1 month
  Describe the rate of margin tumor infiltration
Histological poor outcome predictor rate | 1 month
  Describe the rate of lymphatic, vascular and perineural invasion, histological grade, mean submucosal invasion depth
Radical rescue surgery specimen quality | 1 month
  Describe the quality of Total Mesorectal Excision specimen in terms of mesorectal fascia integrity

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Tovar Perez, MD, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa; Carlos Cerdán Santacruz, PhD, Study Director — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa; Óscar Cano Valderrama, PhD, Study Chair — Complejo Hospitalario Universitario de Vigo; Francisco Jiménez Escovar, PhD, Study Chair — Hospital de Galdakao Usansolo; Blas Flor Lorente, PhD, Study Chair — Hospital Politécnico Universitario la Fe; Javier García Septiem, PhD, Study Chair — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa; Rodrigo Oliva Pérez, PhD, Study Chair — Hospital Alemão Oswaldo Cruz
Locations (1):
- Hospital Universitario de la Princesa, Madrid, Spain

REFERENCES:
- [Derived] Tovar Perez R, Cerdan Santacruz C, Cano-Valderrama O, Jimenez Escovar F, Flor Lorente B, Perez RO, Garcia Septiem J. Local Excision for organ preservation in early REctal cancer with No Adjuvant treatment (LORENA Trial): prospective observational study protocol. Cir Esp (Engl Ed). 2024 Sep;102(9):506-512. doi: 10.1016/j.cireng.2024.04.013. Epub 2024 May 18. PMID 38763491